CLINICAL TRIAL: NCT01346657
Title: The Effect of LipoCol Forte® Capsules on the Pharmacokinetics of Nifedipine After Administering Single-dose Combination to Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yuh-Mou Sue, Department of Internal Medicine, Wanfang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 98030
Record Dates: First submitted 2011-04-27; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Volunteers
Keywords: Nifidipine; red yeast rice; drug-drug interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nifidipine & LipoCol (Experimental): The effect of LipoCol Forte® capsules on the pharmacokinetics of nifedipine after administering single-dose combination in healthy subjects
  Interventions: Drug: Nifidipine & LipoCol

INTERVENTIONS:
Drug: Nifidipine & LipoCol — The effect of LipoCol Forte® capsules on the pharmacokinetics of nifedipine after administering single-dose combination in healthy subjects.

SUMMARY:
The objective of the study is to evaluate the effect of LipoCol Forte® Capsules on the pharmacokinetics of nifedipine after administering single-dose combination to healthy subjects using a 2x2 crossover design.

DETAILED DESCRIPTION:
Healthy subjects were randomly allocated to receive a single dose of either one 5 milgram (mg) nifedipine capsule or one 5 milgram (mg) nifedipine capsule plus one 600 milgram (mg) red yeast rice capsule; after 7-day washout period, they received a single dose of the alternative drug. The subjects were fasted at least 10 hour before dosing. The investigational products were administered with 240 milliliter (mL) of water with the subject in an upright position. The blood samples were collected at prior to the drug administration (T0), and 0.167, 0.333, 0.500, 0.750, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16 and 24 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at the age of 20-40 years old and in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges:Ear body temperature between 35.0-37.5 degree celsius (°C). Systolic blood pressure, 90-140 millimeters of mercury (mm Hg). Diastolic blood pressure, 50-90 millimeters of mercury (mm Hg). Pulse rate, 50-90 beats per minute (bpm). Fasting blood glucose, < 110 milligrams per deciliter (mg/dL).
3. Body weight must be above 50 kilograms (kg) and within -20 to +20% of ideal body weight.
4. Able to sign informed consent prior to study.
5. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. Use of any prescription medication within 14 days prior to dosing.
2. Use of over-the-counter medications or vitamins within 14 days prior to dosing.
3. Significant illness within 2 weeks prior to dosing.
4. Participation in any clinical investigation within 2 months prior to dosing or longer than required by local regulation.
5. Donate or loss more than 500 milliliter(mL) of blood within 3 months prior to dosing.
6. Presence of cardiovascular disease.
7. Presence of gastrointestinal disease.
8. Presence of asthma or lung disease.
9. Presence of liver disease, hepatitis B, hepatitis C or liver injury as indicated by an abnormal liver function profile.
10. Presence of impaired renal function.
11. Presence of neurological disease.
12. Presence of psychiatrical disease.
13. Subject is known for HIV infected.
14. A known hypersensitivity to nifedipine, lovastatin and Chinese Red Yeast Rice or their analogs.
15. History of drug or alcohol abuse within 12 months prior to dosing.
16. Permanent confinement to an institution.
17. Individuals are judged by the investigator or pharmacokineticist to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacokinetic parameters of nifedipine in healthy subjects | 1 week
  Plasma concentrations of nifedipine were detected at following time: (Pre-dose (T0), and 0.167, 0.333, 0.500, 0.750, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16 and 24 hours after oral administration nifedipine capsule with or without red yeast rice capsule (LipoCol)) All pharmacokinetic parameters were determined with nifedipine concentrations by non-compartment methods.

SECONDARY OUTCOMES:
The incidence rate of adverse event | 1 week
  The incidence rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Mou Sue, M.D. Ph.D., Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan